CLINICAL TRIAL: NCT03054376
Title: Impact of Training on Skeletal Muscle Vascular and Metabolic Changes With Limb Immobilization
Brief Title: Vascular Health With Immobilization and Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Johannes Gutenberg University Mainz (Other); University of Leeds (Other); Liverpool John Moores University (Other); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Ylva Hellsten, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ANG-CV- IMMOB
Record Dates: First submitted 2017-02-05; First posted 2017-02-15 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Immobilization, Tonic; Physical Activity
Keywords: Immobilization; Angiogenesis; Skeletal muscle; Exercise training; Vascular function
MeSH Terms: conditions — Immobility Response, Tonic; Motor Activity | interventions — Immobilization; Exercise

STUDY DESIGN:
Intervention Model Description: Parallel randomized to training or no training of non-immobilized leg during immobilization of the other leg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immobilization (Active Comparator): After baseline studies, the subjects will have one leg immobilized by full length plaster for two weeks. During the two weeks, the other leg will not be trained. After the two weeks the subjects will train both legs for four weeks.
  Interventions: Other: Immobilization; Other: Exercise training with both legs
- Training of non-immobilized leg (Active Comparator): After baseline studies, the subjects will have one leg immobilized by full length plaster for two weeks. During the two weeks, the other leg will be trained. After the two weeks the subjects will train both legs for four weeks.
  Interventions: Other: Immobilization; Other: Training with non immobilized leg; Other: Exercise training with both legs

INTERVENTIONS:
Other: Immobilization — Full length cast of one leg R/L randomized
Other: Training with non immobilized leg — Exercise training will be conducted with the non-immobilized leg during the immobilization period of two weeks
  Arms: Training of non-immobilized leg
Other: Exercise training with both legs — Exercise training will be conducted regularly on a cycle ergometer during a four week period

SUMMARY:
The study includes healthy young habitually active subjects. All subjects are subjected to two weeks of immobilization of one leg followed by four weeks of training of both legs. The subjects are randomized to either one-leg training of the non-immobilized leg during the two-week immobilization period or to no training of the non-immobilized leg during the immobilization period. Measures include skeletal muscle morphology, markers of angiogenesis and apoptosis, muscle metabolic markers, vascular function, vascular proteins and performance.

DETAILED DESCRIPTION:
One leg of young healthy subjects will be immoblized for two weeks. Changes in angiogenic proteins and markers of apoptosis in muscle tissue and muscle extracellular fluid will be determined in both legs and in parallel the functional consequences of immobilization will be assessed. Vascular function and vascular proteins will also be determined. In order to understand how the oxidative capacity of the muscle is altered in parallel with changes in capillarization, markers of mitochondria will be measured .Half of the subjects will be randomized to single-leg training during the immobilization period to assess whether simultaneous training reduces the loss of capillaries, muscle function and vascular function in the immobilized leg. After the immobilization period the study participants will train the immobilized leg and the control leg for four weeks by moderate to intense interval cycle training and the same parameteres as during immobilization will be assessed in both legs. The study will also include measurements of circulating compounds and platelets in blood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI <25
* Habitually/moderately physically active

Exclusion Criteria:

* Known chronic medical disorder
* Smoking
* Excessive alcohol intake
* Known genetic/familial predisposition for thrombosis
* Hormonal birth control
* High level strength or endurance training on a regular basis

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Angiogenesis | Change from baseline to after 2 weeks of immobilization
  Skeletal muscle capillarization-comparison between legs
Vascular function | Change from baseline to after 2 weeks of immobilization
  Measurements of skeletal muscle blood flow by ultrasound doppler in response to infusion of vasodilators/constrictors-comparison between legs
Angiogenesis | Change from after immobilization to after 4 weeks of training
  Skeletal muscle capillarization-comparison between legs
Vascular function | Change from after immobilization to after 4 weeks of training
  Measurements of skeletal muscle blood flow by ultrasound doppler in response to infusion of vasodilators/constrictors-comparison between legs

SECONDARY OUTCOMES:
Vascular and metabolic proteins | Change from baseline to after 2 weeks of immobilization and from after immobilization to after 4 weeks of training
  Proteins of importance for vascular function and muscle metabolism measured in muscle biopsy samples, skeletal muscle interstitial fluid and plasma-comparison between legs
Arterial blood pressure | Change from baseline to after 2 weeks of immobilization and from after immobilization to after 4 weeks of training
  Measured by sphygmomanometer and intra-arterially
Knee extensor performance | Change from baseline to after 2 weeks of immobilization and from after immobilization to after 4 weeks of training
  Measurements of maximal power and endurance-comparison between legs
Maximal oxygen uptake | Change from baseline to after 2 weeks of immobilization and from after immobilization to after 4 weeks of training
  Measured by gas analysis during an incremental ergometer cycle protocol
Body composition | Change from baseline to after 2 weeks of immobilization and from after immobilization to after 4 weeks of training
  Measurements by dual energy x-ray absorptiometry
Skin microcirculation | Change from baseline to after 2 weeks of immobilization and from after immobilization to after 4 weeks of training
  Measurements of skin blood flow and morphology and relevant proteins in skin biopsies
Markers of bone metabolism | Change from baseline to after 2 weeks of immobilization and from after immobilization to after 4 weeks of training
  Measurements of bone markers in plasma
Markers of angiogenesis | Change from baseline to after 2 weeks of immobilization and from after immobilization to after 4 weeks of training
  Measurement of angiogenic and apoptotic factors-comparison between legs
Vascular function-non-invasive | Change from baseline to after 2 weeks of immobilization and from after immobilization to after 4 weeks of training
  Measurements of skeletal muscle blood flow at rest, during passive movement, during exercise, after five min of occlusion and during infusion of vasodilators and constrictors-comparison between legs

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gliemann L, Rytter N, Jorgensen TS, Piil P, Carter H, Nyberg M, Grassi M, Daumer M, Hellsten Y. The Impact of Lower Limb Immobilization and Rehabilitation on Angiogenic Proteins and Capillarization in Skeletal Muscle. Med Sci Sports Exerc. 2021 Sep 1;53(9):1797-1806. doi: 10.1249/MSS.0000000000002665. PMID 33787530